CLINICAL TRIAL: NCT00027612
Title: Pilot And Phase II Trial Of Irinotecan And Radiation Followed By Irinotecan And BCNU In Glioblastoma Multiforme Patients
Brief Title: Irinotecan Plus Radiation Therapy Followed By Chemotherapy in Treating Patients With Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N997D; NCCTG-N997D; CDR0000069048 (Registry Identifier: PDQ (Physician Data Query)); NCI-2012-02428 (Registry Identifier: CTRP (Clinical Trials Reporting System)); U10CA025224 (NIH)
Record Dates: First submitted 2001-12-07; First posted 2003-06-17 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — Carmustine; Irinotecan; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- irinotecan + carmustine and radiation (Experimental): Phase II (patients receiving concurrent EIACs or non-EIACs open to accrual as of 3/5/2005): Patients receive irinotecan at the recommended dose, carmustine, and cranial irradiation as in phase I.
  Patients with disease progression are followed every 3 months for 5 years and then annually for up to 10 years.
  Patients taken off study for reasons other than disease progression are followed every 3 months for 1 year, every 6 months for 4 years, and then annually for 5 years.
  Interventions: Drug: carmustine; Drug: irinotecan hydrochloride; Radiation: radiation therapy

INTERVENTIONS:
Drug: carmustine — IV
Drug: irinotecan hydrochloride — IV
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Irinotecan may make the tumor cells more sensitive to radiation therapy.

PURPOSE: This phase I/II trial is studying the side effects of irinotecan given together with radiation therapy followed by irinotecan and carmustine and to see how well it works in treating patients with newly-diagnosed glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety of adjuvant irinotecan when administered concurrently with radiotherapy in patients with newly diagnosed glioblastoma multiforme.
* Determine survival of patients treated with this regimen followed by irinotecan and carmustine.
* Assess the toxic effects of this regimen in these patients.
* Determine whether the dose of irinotecan chosen produces radiosensitizing plasma concentrations of SN-38 in these patients.
* Assess individual variation in responses (toxicity and/or activity), pharmacokinetic parameters, and/or biological correlates due to genetic differences in enzymes involved in transport, metabolism, and/or mechanism of action of irinotecan in these patients treated with this regimen.

OUTLINE: This is a pilot, dose-escalation study of irinotecan. Patients are stratified according to receipt of concurrent enzyme-inducing anticonvulsants (EIACs) (yes vs no).

* Phase I (closed to accrual as of 3/5/2005): Patients receive carmustine IV over 2 hours on day 1 of courses 2-5 and irinotecan IV over 90 minutes (beginning immediately after carmustine infusion) on days 1, 8, 22, and 29 of courses 1-5. Patients also undergo radiotherapy 5 days a week for 6 weeks concurrently with course 1 only. Treatment repeats every 6 weeks for 5 courses in the absence of unacceptable toxicity.

Cohorts of 6 patients receive escalating doses of irinotecan until the recommended dose for phase II is determined. The recommended dose for phase II is defined as the dose at which no more than 2 of 6 patients experience dose-limiting toxicity.

ELIGIBILITY:
* 18 years and older
* Histologically confirmed newly diagnosed grade IV astrocytoma or gliosarcoma
* No oligodendrogliomas/oligoastrocytomas
* Study entry must occur within 8 weeks after surgery
* Performance status - ECOG 0-2
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 130,000/mm^3
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* SGOT ≤ 2 times ULN
* Creatinine ≤ 0.5 mg/dL above ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled infection
* No other concurrent malignant disease except superficial skin cancers
* No other major medical problems
* No prior chemotherapy
* No prior radiotherapy for any tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2002-07; Primary Completion 2006-10 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Survival at 52 weeks | at 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kurt A. Jaeckle, MD, Study Chair — Mayo Clinic

REFERENCES:
- [Result] Jaeckle KA, Ballman KV, Giannini C, Schomberg PJ, Ames MM, Reid JM, McGovern RM, Safgren SL, Galanis E, Uhm JH, Brown PD, Hammack JE, Arusell R, Nikcevich DA, Morton RF, Wender DB, Buckner JC. Phase II NCCTG trial of RT + irinotecan and adjuvant BCNU plus irinotecan for newly diagnosed GBM. J Neurooncol. 2010 Aug;99(1):73-80. doi: 10.1007/s11060-009-0103-2. Epub 2010 Jan 9. PMID 20063115
- [Result] Jaeckle KA, Ballman KV, Schomberg P: N997D: pilot trial of CPT11 during RT followed by CPT11 and BCNU in newly diagnosed glioblastoma (GBM) patients: a North Central Cancer Group (NCCTG) study. [Abstract] J Clin Oncol 23 (Suppl 16): A-1514, 117s, 2005.